CLINICAL TRIAL: NCT06279429
Title: Sucrosomial Iron on Insomnia in Non-dialysis Chronic Kidney Disease Patients With Iron Deficiency Anemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuang Tien General Hospital (Other)
Responsible Party: Principal Investigator, Chun-pai Yang, MD, Chief, Department of Neurology, Kuang Tien General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KTGH11137
Record Dates: First submitted 2024-01-24; First posted 2024-02-28 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: CKD; Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sideral® Sucrosomial Iron (Experimental): The study subjects continued to take Sucrosomial Iron 30mg supplements every day, 2 capsules a day, one 30 minutes after breakfast and dinner, for 12 consecutive weeks. During the study period, none of them used erythropoiesis stimulating agent (ESA).
  Interventions: Dietary Supplement: Sideral® Sucrosomial Iron
- Placebo (Active Comparator): The study subjects continued to take Iron chewable tablet 100mg supplements every day, 2 capsules a day, one 30 minutes after breakfast and dinner, for 12 consecutive weeks. During the study period, none of them used erythropoiesis stimulating agent (ESA).
  Interventions: Dietary Supplement: Iron chewable tablet

INTERVENTIONS:
Dietary Supplement: Sideral® Sucrosomial Iron — Sucrosomial Iron 30mg
  Arms: Sideral® Sucrosomial Iron
Dietary Supplement: Iron chewable tablet — Iron chewable tablet 100mg
  Arms: Placebo

SUMMARY:
Insomnia or sleep disturbance is a common disorder in patients with chronic kidney disease (CKD), but is often unrecognized and undertreated. It is known that sleep disorders may indirectly cause a variety of diseases and affect quality of life. The most common sleep disorders that occur in CKD are insomnia, excessive daytime sleepiness, obstructive or central sleep apnea (SA), and sleep disorders. This study evaluates the effectiveness and safety of Sideral® Sucrosomial Iron and iron chewable tablets 100mg commonly used in health insurance on sleep disorders in patients with CKD and iron deficiency anemia.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 20-80.
2. Chronic kidney disease (CKD) patients.
3. Iron deficiency anemia (male haemoglobin (Hb) ≤13 g/dL; female haemoglobin (Hb) ≤12 g/dL, ferritin ≤100 ng/mL, transferrin saturation ≤25%).
4. Patients diagnosed as chronic insomnia by doctors according to international classification of sleep disorders-third edition (ICSD-3).
5. Subjects who voluntarily participate in the trial plan and complete the consent form after explanation by doctors or project personnel.

Exclusion Criteria:

1. Patients taking iron supplements.
2. Patients with non-chronic insomnia.
3. Patients with alcoholism within one year.
4. People with other serious diseases.
5. Pregnant women or women who are still breastfeeding.
6. Those who are unable to cooperate with the test progress.
7. Patients with autoimmune abnormalities (ex. inflammatory bowel disease).
8. People with non-iron deficiency anemia (ex. thalassemia).
9. Those who are taking sleeping pills or sedatives.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | week 0, 12
  A sleep-related questionnaire, ranging from 0 to 28, where higher scores indicate more acute symptoms of insomnia.
Pittsburgh Sleep Quality Index (PSQI) | week 0, 12
  A sleep-related questionnaire, ranging from 0 to 21 with the higher total score indicating worse sleep quality.
Epworth sleepiness Scale (ESS) | week 0, 12
  A sleep-related questionnaire, ranging from 0 to 24. Scores from 0 to 10 reflect normal levels of daytime sleepiness, and scores over 10 are considered to reflect excessive daytime sleepiness.
Hemoglobin | week 0, 12
  Concentration of serum hemoglobin
Ferritin | week 0, 12
  Concentration of serum ferritin
Serum Iron | week 0, 12
  Concentration of serum Iron
Transferrin Saturation | week 0, 12
  Concentration of serum transferrin Saturation
Erythrocyte sedimentation rate | week 0, 12
  Concentration of serum erythrocyte sedimentation rate

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Pai Yang, MD, Principal Investigator — Chief, Department of Neurology
Locations (1):
- Kuang Tien General Hospital, Taichung, Taiwan